CLINICAL TRIAL: NCT05422144
Title: BIAKOS Antimicrobial Wound Cleanser and BIAKOS Antimicrobial Wound Gel: Providing Biofilm Prevention and Treatment Through Continuum of Care
Brief Title: Cleanser for Acute Wounds
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: That aim was forfeited due to enrollment challenges and lack of remaining funding to accomplish.
Sponsor: Rochal Industries LLC (Industry)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other); MicroGenDX (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTEC-20-02-Multi-Topic-017
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Wound
Keywords: Traumatic Wounds; Biofilm; Antimicrobial; Sepsis; Infection; Wound
MeSH Terms: conditions — Sepsis; Infections; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Antimicrobial Skin & Wound Cleanser and Antimicrobial Wound gel will be subsequently administered to the wound during the 28 day study duration.
  Interventions: Device: Antimicrobial Skin & Wound Cleanser (AWC); Device: Antimicrobial Wound Gel (AWG)

INTERVENTIONS:
Device: Antimicrobial Skin & Wound Cleanser (AWC) — BIAKŌS™ Antimicrobial Skin & Wound Cleanser helps in the mechanical removal of debris and foreign material from the skin, wound, or application site. BIAKŌS™ Antimicrobial Skin and Wound Cleanser is a pure, colorless, isotonic cleanser that is safe. The preservative, polyhexamethylene biguanide (PHMB), at a concentration of 0.1% w/w is added to the product to inhibit the growth of microorganisms such as Staphylococcus aureus, Staphylococcus epidermidis, Pseudomonas aeruginosa, Escherichia coli, antibiotic resistant Methicillin Resistant Staphylococcus aureus (MRSA). and fungus Candida albicans within the product.
  Other Names: BIAKŌS Antimicrobial Skin & Wound Cleanser; AWC
Device: Antimicrobial Wound Gel (AWG) — BIAKŌS Antimicrobial Wound Gel provides a moist environment to wound surfaces. BIAKŌS Antimicrobial Wound Gel is a safe and gentle colorless gel. The gel provides preservative properties through the antimicrobial polyhexamethylene biguanide (PHMB).
  BIAKŌS Antimicrobial Wound Gel:
  * Resists microbial colonization within the gel during shelf storage.
  * Provides an amorphous gel covering.
  * Facilitates autolytic debridement through a moist wound environment. Wounds experience some level of autolytic debridement in which the body's own enzymes breakdown necrotic tissue.
  Other Names: BIAKŌS Antimicrobial Wound Gel; AWG

SUMMARY:
The proposed study will be a prospective trial of management of acute traumatic wounds (less than 24 hours from injury and without previous intervention aside from a dressing for coverage). The study design involves a prospective single arm, 35 subject study that analyzes the effect of the subsequent application of a novel wound cleanser and wound gel on subjects' acute traumatic wounds and the respective microbial loads over a 28 day study duration.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 89 years old.
* Patients receiving care in the ED/trauma bay or admitted to Brooke Army Medical Center (BAMC) from the ED or trauma bay.
* At least one wound area must measure equal to or greater than 2cm^2 to include partial or full thickness tears.
* Wound sustained less than 48-hours from time of enrollment.
* The wound must be untreated/open beyond bedside stabilization such as irrigation and debridement (i.e., no stitches, steristrips, dermabond, OR washouts, etc).
* Capable of providing informed written consent by self or through Legally Authorized Representative (LAR).
* Ability to read/speak English (participant and/ or LAR).

Exclusion Criteria:

* Ages less than 18 or greater than 89 years old.
* Patients not receiving care in the ED/trauma bay or admitted to BAMC through the ED or trauma bay.
* Wound area less than 2 cm2.
* Wound sustained greater than 48-hours from the time of enrollment.
* Wounds that have been closed/repaired at the time of screening (i.e. stitches, steristrips, dermabond, washouts in the OR, etc.) or anytime during the study duration.
* Not capable of providing informed written consent by self or through LAR.
* Non-English reading and speaking (participant and/or LAR).
* Have received more than one dose of antibiotics prior to enrollment or during the study duration.
* Suspected or confirmed signs/symptoms of active wound infection or gangrene.
* Patients with osteomyelitis.
* Wounds with exposed tendons, ligaments, or bone.
* Patients undergoing active renal dialysis.
* Patients receiving (within 30 days of enrollment) or scheduled to receive a medication or treatment which is known to negatively affect wound healing such as systemic steroids (i.e. continuous prednisone), immunosuppressive therapy, chemotherapy, autoimmune disease therapy, cytostatic therapy, vascular surgery, angioplasty, or thrombolysis.
* Pregnant, breastfeeding, or women of childbearing potential who do not agree to use an effective form of contraception during their participation in the study.
* Participation in another investigational device, drug, or biological trial that may interfere with results within 30 days of screening.
* Anyone deemed by the PI to be unlikely to comply with all study procedures.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Microbial Load | 28 days
  As indicated semi-quantitatively by MicroGenDx/ Research and Testing Labs LLC (RTL) swab collection and qualitatively by visual assessments and MolecuLight i:X images.

SECONDARY OUTCOMES:
Wound Healing Rates | 28 days
  % reduction in wound bed size over time as determined by wound measurement and Bates-Jensen Wound Assessment Tool

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Mcmahon, Masters, Principal Investigator — Rochal Industires
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The data collected for this study will remain within the access of the study team and collaborators only. The same study team will utilize this data to compare with a retrospective study to serve as the control comparison for this study. This data will not be shared with other researchers.

REFERENCES:
- [Background] Army, O. of T. S. G. U. S. Infections. Emergency War Surgery, Fourth United States Revision (2013).
- [Background] Black CE, Costerton JW. Current concepts regarding the effect of wound microbial ecology and biofilms on wound healing. Surg Clin North Am. 2010 Dec;90(6):1147-60. doi: 10.1016/j.suc.2010.08.009. PMID 21074033
- [Background] Bowler PG, Duerden BI, Armstrong DG. Wound microbiology and associated approaches to wound management. Clin Microbiol Rev. 2001 Apr;14(2):244-69. doi: 10.1128/CMR.14.2.244-269.2001. PMID 11292638
- [Background] Church D, Elsayed S, Reid O, Winston B, Lindsay R. Burn wound infections. Clin Microbiol Rev. 2006 Apr;19(2):403-34. doi: 10.1128/CMR.19.2.403-434.2006. PMID 16614255
- [Background] Percival SL, Hill KE, Williams DW, Hooper SJ, Thomas DW, Costerton JW. A review of the scientific evidence for biofilms in wounds. Wound Repair Regen. 2012 Sep-Oct;20(5):647-57. doi: 10.1111/j.1524-475X.2012.00836.x. PMID 22985037
- [Background] Donlan RM, Costerton JW. Biofilms: survival mechanisms of clinically relevant microorganisms. Clin Microbiol Rev. 2002 Apr;15(2):167-93. doi: 10.1128/CMR.15.2.167-193.2002. PMID 11932229
- [Background] Hoiby N, Bjarnsholt T, Givskov M, Molin S, Ciofu O. Antibiotic resistance of bacterial biofilms. Int J Antimicrob Agents. 2010 Apr;35(4):322-32. doi: 10.1016/j.ijantimicag.2009.12.011. Epub 2010 Feb 10. PMID 20149602
- [Background] Leid JG, Willson CJ, Shirtliff ME, Hassett DJ, Parsek MR, Jeffers AK. The exopolysaccharide alginate protects Pseudomonas aeruginosa biofilm bacteria from IFN-gamma-mediated macrophage killing. J Immunol. 2005 Dec 1;175(11):7512-8. doi: 10.4049/jimmunol.175.11.7512. PMID 16301659
- [Background] Stewart PS, Costerton JW. Antibiotic resistance of bacteria in biofilms. Lancet. 2001 Jul 14;358(9276):135-8. doi: 10.1016/s0140-6736(01)05321-1. PMID 11463434
- [Background] Gutierrez D, Hidalgo-Cantabrana C, Rodriguez A, Garcia P, Ruas-Madiedo P. Monitoring in Real Time the Formation and Removal of Biofilms from Clinical Related Pathogens Using an Impedance-Based Technology. PLoS One. 2016 Oct 3;11(10):e0163966. doi: 10.1371/journal.pone.0163966. eCollection 2016. PMID 27695058
- [Background] Wolcott RD, Rhoads DD, Bennett ME, Wolcott BM, Gogokhia L, Costerton JW, Dowd SE. Chronic wounds and the medical biofilm paradigm. J Wound Care. 2010 Feb;19(2):45-6, 48-50, 52-3. doi: 10.12968/jowc.2010.19.2.46966. PMID 20216488
- [Background] Rasmussen TE, Baer DG, Remick KN, Ludwig GV. Combat casualty care research for the multidomain battlefield. J Trauma Acute Care Surg. 2017 Jul;83(1 Suppl 1):S1-S3. doi: 10.1097/TA.0000000000001469. No abstract available. PMID 28628599
- [Background] Harris C, Bates-Jensen B, Parslow N, Raizman R, Singh M, Ketchen R. Bates-Jensen wound assessment tool: pictorial guide validation project. J Wound Ostomy Continence Nurs. 2010 May-Jun;37(3):253-9. doi: 10.1097/WON.0b013e3181d73aab. PMID 20386331
- [Background] Raizman R, Dunham D, Lindvere-Teene L, Jones LM, Tapang K, Linden R, Rennie MY. Use of a bacterial fluorescence imaging device: wound measurement, bacterial detection and targeted debridement. J Wound Care. 2019 Dec 2;28(12):824-834. doi: 10.12968/jowc.2019.28.12.824. PMID 31825778
- [Background] Guidance for Industry Chronic Cutaneous Ulcer and Burn Wounds - Developing Products for Treatment. U.S. Department of Health and Human Services Food and Drug Administration Center for Drug Evaluation and Research (CDER) Center for Biologics Evaluation and Research (CBER) Center for Devices and Radiological Health (CDRH) June 2006 Clinical/Medical. https://www.fda.gov/media/71278/download
- [Background] Fleming TR. One-sample multiple testing procedure for phase II clinical trials. Biometrics. 1982 Mar;38(1):143-51. PMID 7082756
- [Background] Schultz JR, Nichol FR, Elfring GL, Weed SD. Multiple-stage procedures for drug screening. Biometrics. 1973 Jun;29(2):293-300. No abstract available. PMID 4709516
- [Background] Jennison, C. & Turnbull, B., Group Sequential Methods with Applications to Clinical Trials. (Chapman & Hall/CRC, 2000).
- [Background] Belmont PJ, Schoenfeld AJ, Goodman G. Epidemiology of combat wounds in Operation Iraqi Freedom and Operation Enduring Freedom: orthopaedic burden of disease. J Surg Orthop Adv. 2010 Spring;19(1):2-7. PMID 20370999
- [Background] Geiling J, Rosen JM, Edwards RD. Medical costs of war in 2035: long-term care challenges for veterans of Iraq and Afghanistan. Mil Med. 2012 Nov;177(11):1235-44. doi: 10.7205/milmed-d-12-00031. PMID 23198496
- [Background] Mende K, Stewart L, Shaikh F, Bradley W, Lu D, Krauss MR, Greenberg L, Yu Q, Blyth DM, Whitman TJ, Petfield JL, Tribble DR. Microbiology of combat-related extremity wounds: Trauma Infectious Disease Outcomes Study. Diagn Microbiol Infect Dis. 2019 Jun;94(2):173-179. doi: 10.1016/j.diagmicrobio.2018.12.008. Epub 2018 Dec 29. PMID 30691724